CLINICAL TRIAL: NCT02813681
Title: A Prospective Randomized Clinical Trial to Study the Effect of Pre-Epidural Ultrasound Examination on Epidural Insertion Site Pressure Sensitivity in Parturient
Brief Title: Ultrasound-Guided Landmark and Epidural Site Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-0110
Record Dates: First submitted 2016-06-16; First posted 2016-06-27 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2016-06

CONDITIONS: Back Pain; Epidural Analgesia, Obstetric
Keywords: Acute Pain; ultrasonography
MeSH Terms: conditions — Back Pain; Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- US-epidural SVD (Active Comparator): US-epidural SVD group - participants who received US examination prior to epidural placement. The purpose of this group is to determine if US derived landmarks reduce pressure sensitivity
  Interventions: Procedure: US-epidural SVD
- (US sham- epidural SVD) (Sham Comparator): US sham- epidural SVD group- participants who received US examination process but with the monitor turned off.
  Interventions: Procedure: US sham- epidural SVD
- SVD without an Epidural (Placebo Comparator): Spontaneous vaginal delivery without an Epidural group The purpose of the control group is to serve as a baseline.
  Interventions: Procedure: Spontaneous vaginal delivery without an Epidural

INTERVENTIONS:
Procedure: US-epidural SVD — participants who received US examination prior to epidural placement. The purpose of this group is to determine if US derived landmarks reduce pressure sensitivity.
  Arms: US-epidural SVD
Procedure: US sham- epidural SVD — participants who received US examination process but with the monitor turned off. The purpose of this group is to determine if the standard of care epidural placement technique will increase pressure sensitivity at the insertion site. The purpose of this group will also be to reduce the placebo effect from the US exam and to maintain blinding of the patient to their group status (US epidural or US sham epidural).
  Arms: (US sham- epidural SVD)
Procedure: Spontaneous vaginal delivery without an Epidural — Spontaneous vaginal delivery without an Epidural The purpose of the control group is to serve as a baseline (or a measure of normal). The control participant's measurement will be compared to those that did receive treatments (either epidural alone or ultrasound and epidural). This information will tell the investigator how many women have back pain after spontaneous vaginal delivery. Participant must meet the inclusion requirements and not meet any of the exclusion requirements
  Arms: SVD without an Epidural

SUMMARY:
Historically, women who have chronic back pain after pregnancy have attributed the cause to the epidural procedure. While many studies have shown no greater incidence of generalized post-partum back pain in those who received an epidural, no studies have measured localized pressure sensitivity at the epidural insertion site. Short-term pressure sensitivity might limit patient's mobility and activities in the post-partum period. Understanding the factors that increase insertion site pressure sensitivity will allow the investigators to modify epidural placement technique in order to minimize this effect.

DETAILED DESCRIPTION:
Few studies have examined how epidural placement changes localized sensation at the epidural insertion site. This study will be the first study to quantitatively measure sensation at the epidural insertion site. The investigator will assess localized pressure sensitivity with an algometer. An algometer is a hand-held device commonly used by neurologist to detect sensory deficits and measures the pressure sensitivity threshold in a 1-cm diameter circular area. Ultrasound (US) pre-procedural examination provides more accurate landmarks for the placement of epidural catheters. The investigator will determine if an US examination prior to epidural placement reduces localized pressure sensitivity. The investigator will also determine if there are correlations between the participants characteristics and/or comorbidities and increased pressure sensitivity at the insertion site.

ELIGIBILITY:
Inclusion Criteria:

* pregnant with term (37 - 41 weeks) singleton gestation
* active labor
* history of normal pregnancy
* request an epidural
* age between 18 - 35 years old
* able to understand the protocol and provide voluntary, written, informed consent.

Exclusion Criteria:

* history of spinal surgery
* scoliosis
* epidural or spinal placement within the last 5 days
* neuropathic pain disorders
* chronic opioid use
* Texas Department of Criminal Justice patient
* placental percreta
* placental increta
* placenta accreta
* preeclampsia
* eclampsia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Wilkes, Principal Investigator — UTMB

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- US-epidural SVD: Group 1: (US-epidural SVD) - participants who received US examination prior to epidural placement. The purpose of this group is to determine if US derived landmarks reduce pressure sensitivity
  US-epidural SVD: participants who received US examination prior to epidural placement. The purpose of this group is to determine if US derived landmarks reduce pressure sensitivity.
  Algometer: Wagner FPX series manual algometer will be used to assess pain pressure threshold.
- (US Sham- Epidural SVD): Group 2: (US sham- epidural SVD) - participants who received US examination process but with the monitor turned off. The purpose of this group is to determine if the standard of care epidural placement technique will increase pressure sensitivity at the insertion site. The purpose of this group will also be to reduce the placebo effect from the US exam and to maintain blinding of the participant to their group status (US epidural or US sham epidural).
  US sham- epidural SVD: participants who received US examination process but with the monitor turned off. The purpose of this group is to determine if the standard of care epidural placement technique will increase pressure sensitivity at the insertion site. The purpose of this group will also be to reduce the placebo effect from the US exam and to maintain blinding of the patient to their group status (US epidural or US sham epidural).
  Algometer: Wagner FPX series manual algometer will be used to assess pain pressure threshold.
- Spontaneous Vaginal Delivery Without an Epidural: Group 5: Spontaneous vaginal delivery without an Epidural The purpose of the control group is to serve as a baseline (or a measure of normal). The control participant's measurement will be compared to those that did receive treatments (either epidural alone or ultrasound and epidural).
  Spontaneous vaginal delivery without an Epidural: Spontaneous vaginal delivery without an Epidural The purpose of the control group is to serve as a baseline (or a measure of normal). The control participant's measurement will be compared to those that did receive treatments (either epidural alone or ultrasound and epidural). This information will tell the investigator how many women have back pain after spontaneous vaginal delivery. Participant must meet the inclusion requirements and not meet any of the exclusion requirements
  Algometer: Wagner FPX series manual algometer will be used to assess pain pressure threshold.
Period: Overall Study
Arm/Group | US-epidural SVD | (US Sham- Epidural SVD) | Spontaneous Vaginal Delivery Without an Epidural
Started | 27 | 34 | 19
Completed | 22 | 28 | 19
Not Completed | 5 | 6 | 0
Not completed — Physician Decision | 5 | 5 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants who elected to get an epidural proceed to spontaneous vaginal surgery
Groups:
- US-epidural SVD: US-epidural SVD group- participants who received US examination prior to epidural placement. The purpose of this group is to determine if US derived landmarks reduce pressure sensitivity
  US-epidural SVD: participants who received US examination prior to epidural placement. The purpose of this group is to determine if US derived landmarks reduce pressure sensitivity.
  Algometer: Wagner FPX series manual algometer will be used to assess pain pressure threshold.
- (US Sham- Epidural SVD): US sham- epidural SVD group - participants who received US examination process but with the monitor turned off. The purpose of this group is to determine if the standard of care epidural placement technique will increase pressure sensitivity at the insertion site. The purpose of this group will also be to reduce the placebo effect from the US exam and to maintain blinding of the participant to their group status (US epidural or US sham epidural).
  US sham- epidural SVD: participants who received US examination process but with the monitor turned off. The purpose of this group is to determine if the standard of care epidural placement technique will increase pressure sensitivity at the insertion site. The purpose of this group will also be to reduce the placebo effect from the US exam and to maintain blinding of the patient to their group status (US epidural or US sham epidural).
  Algometer: Wagner FPX series manual algometer will be used to assess pain pressure threshold.
- Spontaneous Vaginal Delivery Without an Epidural: Spontaneous vaginal delivery without an Epidural group The purpose of the control group is to serve as a baseline (or a measure of normal). The control participant's measurement will be compared to those that did receive treatments (either epidural alone or ultrasound and epidural).
  The purpose of the control group is to serve as a baseline (or a measure of normal). The control participant's measurement will be compared to those that did receive treatments (either epidural alone or ultrasound and epidural). This information will tell the investigator how many women have back pain after spontaneous vaginal delivery. Participant must meet the inclusion requirements and not meet
- Total: Total of all reporting groups
Arm/Group | US-epidural SVD | (US Sham- Epidural SVD) | Spontaneous Vaginal Delivery Without an Epidural | Total
Number analyzed (Participants) | 22 | 28 | 19 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 28 | 19 | 69
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (1.3) | 26.3 (1.2) | 26.6 (1) | 26.4 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 19 | 69
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 28 | 19 | 69
body mass index [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (1) | 26.3 (1.2) | 26.6 (1) | 28 (1.1)
number of prior births [Mean (Standard Deviation); unit: births] | 2.2 (0.2) | 3 (0.4) | 3 (1.5) | 2.7 (0.3)
length of labor [Mean (Standard Deviation); unit: hours] | 10.9 (1.3) | 12 (1.4) | 8 (0.9) | 10.3 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Epidural Pressure Sensitivity at Level of Epidural Insertion
Description: pressure sensitivity at level of epidural insertion will be measured with an algometer (Newtons)
Time Frame: Epidural pressure sensitivity was monitored 10 minutes prior to epidural insertion and then for 10 minutes on each day after epidural removal for 3 days.
Population: pressure sensitivity at level of epidural insertion will be measured at epidural insertion site level.
Measure: Mean (Standard Error); unit: force (newtons/cm^2)
Groups:
- US-epidural SVD: US-epidural SVD group - participants who received US examination prior to epidural placement. The purpose of this group is to determine if US derived landmarks reduce pressure sensitivity
  US-epidural SVD: participants who received US examination prior to epidural placement. The purpose of this group is to determine if US derived landmarks reduce pressure sensitivity.
  Algometer: Wagner FPX series manual algometer will be used to assess pain pressure threshold.
- (US Sham- Epidural SVD): US sham- epidural SVD group- participants who received US examination process but with the monitor turned off. The purpose of this group is to determine if the standard of care epidural placement technique will increase pressure sensitivity at the insertion site. The purpose of this group will also be to reduce the placebo effect from the US exam and to maintain blinding of the participant to their group status (US epidural or US sham epidural).
  US sham- epidural SVD: participants who received US examination process but with the monitor turned off. The purpose of this group is to determine if the standard of care epidural placement technique will increase pressure sensitivity at the insertion site. The purpose of this group will also be to reduce the placebo effect from the US exam and to maintain blinding of the patient to their group status (US epidural or US sham epidural).
  Algometer: Wagner FPX series manual algometer will be used to assess pain pressure threshold.
- Spontaneous Vaginal Delivery Without an Epidural: Spontaneous vaginal delivery without an Epidural group The purpose of the control group is to serve as a baseline (or a measure of normal). The control participant's measurement will be compared to those that did receive treatments (either epidural alone or ultrasound and epidural).
  Spontaneous vaginal delivery without an Epidural: Spontaneous vaginal delivery without an Epidural The purpose of the control group is to serve as a baseline (or a measure of normal). The control participant's measurement will be compared to those that did receive treatments (either epidural alone or ultrasound and epidural). This information will tell the investigator how many women have back pain after spontaneous vaginal delivery. Participant must meet the inclusion requirements and not meet any of the exclusion requirements
  Algometer: Wagner FPX series manual algometer will be used to assess pain pressure threshold.
Arm/Group | US-epidural SVD | (US Sham- Epidural SVD) | Spontaneous Vaginal Delivery Without an Epidural
Number analyzed (Participants) | 22 | 28 | 19
force (newtons/cm^2) | 26.8 (3.2) | 26.8 (2.4) | 47.6 (2.3)

2. Secondary Outcome: Induction Medication
Description: The investigator will review the chart to see if the participant used of induction medication (answer yes will be recorded)
Time Frame: The chart review will determine the use of induction medication immediately prior to the epidural placement
Measure: Count of Participants; unit: Participants
Arm/Group | US-epidural SVD | (US Sham- Epidural SVD) | Spontaneous Vaginal Delivery Without an Epidural
Number analyzed (Participants) | 22 | 28 | 19
Participants | 22 | 28 | 17

3. Secondary Outcome: Opioid Use During Labor
Description: The investigator will review the chart to see if the participant required opioids during labor (yes will be recorded)
Time Frame: A chart review of systemic opioids given to participant when the epidural is removed
Measure: Count of Participants; unit: Participants
Arm/Group | US-epidural SVD | (US Sham- Epidural SVD) | Spontaneous Vaginal Delivery Without an Epidural
Number analyzed (Participants) | 22 | 28 | 19
Participants | 6 | 9 | 9

4. Secondary Outcome: Short-term Back Pain
Description: The investigator will ask the participant if they have had back pain lasting longer than one week during pregnancy? (yes answer will be recorded)
Time Frame: Participants will be asked if they have had back pain for longer than a week immediately prior to epidural placement
Measure: Count of Participants; unit: Participants
Arm/Group | US-epidural SVD | (US Sham- Epidural SVD) | Spontaneous Vaginal Delivery Without an Epidural
Number analyzed (Participants) | 22 | 28 | 19
Participants | 4 | 7 | 7

5. Secondary Outcome: Number of Needle Repositions
Description: The investigator will count the number epidural needle repositions during the epidural placement (whole number)
Time Frame: The number of needle reposition will be counted during epidural placement.
Population: The SVD without an epidural is not included in this analysis because this group did not get an epidural and therefore will not have needle repositions.
Measure: Mean (Standard Error); unit: number of needle repositions
Arm/Group | US-epidural SVD | (US Sham- Epidural SVD)
Number analyzed (Participants) | 22 | 28
number of needle repositions | 0.8 (0.1) | 2.2 (0.3)

6. Secondary Outcome: Number of Needle Insertions
Description: The investigator will count the number epidural needle insertions during the epidural placement (whole number)
Time Frame: The number of needle insertions will be counted during epidural placement.
Measure: Mean (Standard Error); unit: number of needle insertions
Arm/Group | US-epidural SVD | (US Sham- Epidural SVD)
Number analyzed (Participants) | 22 | 28
number of needle insertions | 0.1 (.01) | .8 (.1)

ADVERSE EVENTS:
Groups:
- Spontaneous Vaginal Delivery Without an Epidural: Group 5: Spontaneous vaginal delivery without an Epidural The purpose of the control group is to serve as a baseline (or a measure of normal). The control participant's measurement will be compared to those that did receive treatments (either epidural alone or ultrasound and epidural).
  The purpose of the control group is to serve as a baseline (or a measure of normal). The control participant's measurement will be compared to those that did receive treatments (either epidural alone or ultrasound and epidural). This information will tell the investigator how many women have back pain after spontaneous vaginal delivery. Participant must meet the inclusion requirements and not meet
Arm/Group | US-epidural SVD | (US Sham- Epidural SVD) | Spontaneous Vaginal Delivery Without an Epidural
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/28 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/28 | 0/19
Other Adverse Events (participants affected / at risk) | 0/22 | 0/28 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No